CLINICAL TRIAL: NCT00513448
Title: Comparing Individualized Rehabilitation to a Group Wellness Intervention for Persons With Multiple Sclerosis
Brief Title: Promoting Physical Activity for Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0311M53442
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-08

CONDITIONS: Multiple Sclerosis
Keywords: Chronic Disabling Condition; Comparative Evaluation; Physical Activity; Physical Therapy; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Group wellness intervention
Other: Individualized physical rehabilitation

SUMMARY:
The purpose of this study was to determine whether a group wellness intervention or individualized physical rehabilitation was more effective in improving health and physical activity in persons with multiple sclerosis.

DETAILED DESCRIPTION:
Evidence from this study shows that both interventions were effective in improving health and physical activity in persons with multiple sclerosis. The results also show that participants may benefit more physically from individualized physical rehabilitation and more mentally from group wellness interventions. Interventions that combine individualized therapeutic exercise with group health education might be most effective for persons with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* A physician-confirmed diagnosis of MS
* Between the ages of 18 to 75 years
* Ability to ambulate 25 meters with or without the use of an adaptive aide

Exclusion Criteria:

* Pregnant
* Cardiovascular disease
* Had fallen more than twice in the past month
* Significant cognitive deficits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-04; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale SF-36 Mental Health Inventory | 16 weeks

SECONDARY OUTCOMES:
Physical assessments | 16-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Plow, PhD, Principal Investigator — Brown University
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States